CLINICAL TRIAL: NCT05523518
Title: Which Technique is Effective in Reducing the Pain of Peripheral Intravenous Catheterization in Pediatric Patients, Infra-Red Light or Buzzy®?
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Uludag University (Other)
Responsible Party: Principal Investigator, Dilek Yilmaz, PhD, Bursa Uludag University, Department of Nursing, Uludag University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 2022-10/22
Record Dates: First submitted 2022-08-28; First posted 2022-08-31 (Actual); Last update posted 2022-08-31 (Actual); Status verified 2022-08

CONDITIONS: Pain Management
Keywords: pain control; nonpharmacological method; AccuVein®; Buzzy®; pediatric patients; peripheral intravenous catheterization
MeSH Terms: conditions — Agnosia

STUDY DESIGN:
Who Masked: Investigator
Masking Description: The intervention and measurements were carried out by the researcher
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (3):
- The Buzzy® group (Experimental): From one minute before the location of the catheter and until the end of the procedure, the researchers will place the Buzzy® device approximately 5cm above the area where the procedure will take place, with its wings under it. The gel in its wings will have been previously frozen solid in a refrigerator. In this way, vibration and cold will be applied, and immediately afterwards, vein entry will be performed. (For the children's safety, a piece of thin sterile gauze will be placed on the area in order to prevent direct contact between the ice wings and the skin.)
  Interventions: Device: The Buzzy®
- the AccuVein® group (Experimental): In this group, the veins in the area where the entry is to be performed will be visualized with the AccuVein® infrared vein visualization device, and the standard catheter implementation will be performed in the vein which is decided on for entry.
  Interventions: Device: The AccuVein®
- The control group (No Intervention): With the pediatric patients in the control group, no intervention will be performed before or during the procedure, and routine IV catheterization will be carried out without the use of any device.

INTERVENTIONS:
Device: The Buzzy® — From one minute before the location of the catheter and until the end of the procedure, the researchers will place the Buzzy® device approximately 5cm above the area where the procedure will take place, with its wings under it. The gel in its wings will have been previously frozen solid in a refrigerator. In this way, vibration and cold will be applied, and immediately afterwards, vein entry will be performed. (For the children's safety, a piece of thin sterile gauze will be placed on the area in order to prevent direct contact between the ice wings and the skin.)
  Arms: The Buzzy® group
Device: The AccuVein® — In this group, the veins in the area where the entry is to be performed will be visualized with the AccuVein® infrared vein visualization device, and the standard catheter implementation will be performed in the vein which is decided on for entry.
  Arms: the AccuVein® group

SUMMARY:
The aim of this study is to examine the effect on the pain developing from peripheral intravenous catheterization (IV) in pediatric patients of an infra-red vein visualization device, AccuVein®, and Buzzy®, which can simultaneously produce vibration and cold.

The research is planned as a prospective, randomized controlled study with an experimental design. Research data collection will be conducted at the Pediatric Emergency Service of the Health Research and Application Center of Bursa Uludağ University. The research sample will consist of children aged 7-12 years who attend the Pediatric Emergency Service of the Health Research and Application Center of Bursa Uludağ University for diagnosis or treatment, who have been ordered a peripheral intravenous catheter for intravenous treatment by a doctor, and whose participation is voluntarily accepted by themselves and their parents. It was calculated as a result of power analysis that the minimum sample size is 90 child patients, with 30 in each group, to reach an 80% power level, accepting a type I error level of 5%. Pediatric patients who fit the inclusion criteria of the study will be assigned to implementation and control groups with the use of a computer-generated randomization list, according to their age and gender.

An Individual Data Collection Form and the Facial Expressions Pain Rating Scale will be used to collect data by face to face interview.

Peripheral intravenous catheterization will be implemented on the veins of either the right or the left arm. The procedural steps of the standard vein entry protocol will be followed with all of the children in the implementation and control groups.

In addition to the standard vein entry protocol, the following interventions will be conducted with the pediatric patients in the implementation groups.

Peripheral intravenous catheterization with pediatric patients in the Buzzy® group: From one minute before the location of the catheter and until the end of the procedure, the researchers will place the Buzzy® device approximately 5cm above the area where the procedure will take place, with its wings under it. The gel in its wings will have been previously frozen solid in a refrigerator. In this way, vibration and cold will be applied, and immediately afterwards, vein entry will be performed. (For the children's safety, a piece of thin sterile gauze will be placed on the area in order to prevent direct contact between the ice wings and the skin.)

Peripheral intravenous catheterization with pediatric patients in the AccuVein® group: In this group, the veins in the area where the entry is to be performed will be visualized with the AccuVein® infrared vein visualization device, and the standard catheter implementation will be performed in the vein which is decided on for entry.

Peripheral intravenous catheterization with pediatric patients in the control group: With the pediatric patients in the control group, no intervention will be performed before or during the procedure, and routine IV catheterization will be carried out without the use of any device.

Immediately after the procedure has been performed, an assistant researcher who is unaware of the catheterization method used will ask the children of all groups to assess their pain levels with the Facial Expressions Pain Rating Scale, and the scores indicated will be recorded on the data collection form. While the study is being conducted, the necessary measures will be taken to prevent the children included in the study from influencing each other, such as not allowing them to see the method applied to the other children.

DETAILED DESCRIPTION:
The aim of this study is to examine the effect on the pain developing from peripheral intravenous catheterization (IV) in pediatric patients of an infra-red vein visualization device, AccuVein®, and Buzzy®, which can simultaneously produce vibration and cold.

The research is planned as a prospective, randomized controlled study with an experimental design. Research data collection will be conducted at the Pediatric Emergency Service of the Health Research and Application Center of Bursa Uludağ University. The research sample will consist of children aged 7-12 years who attend the Pediatric Emergency Service of the Health Research and Application Center of Bursa Uludağ University for diagnosis or treatment, who have been ordered a peripheral intravenous catheter for intravenous treatment by a doctor, and whose participation is voluntarily accepted by themselves and their parents.

The size of the study sample was statistically determined with the program G*Power 3.1.7. It was calculated as a result of power analysis that the minimum sample size is 90 child patients, with 30 in each group, to reach an 80% power level, accepting a type I error level of 5%. Pediatric patients who fit the inclusion criteria of the study will be assigned to implementation and control groups with the use of a computer-generated randomization list, according to their age and gender. That is, the study group in which the children are placed will be determined by a randomization method according to a randomization list.

An Individual Data Collection Form and the Facial Expressions Pain Rating Scale will be used to collect data by face to face interview.

Individual Data Collection Form: This form will have questions on the children's age, gender, height, weight, the vein where the catheter is located (left or right), and the duration of catheterization.

Facial Expressions Pain Rating Scale: This scale depends on various different facial expressions depicted visually. It is used in clinical pediatric implementations to measure pain severity. The expression of no pain is generally shown with a smiling face, and the worst pain with a crying face.

The pediatric patients to be included in the study and their parents will be informed about the research, and oral approval will be obtained from the children and oral and written approval will be obtained from their parents. After securing their voluntary participation, the children will be assigned to implementation and control groups. After that, the children's descriptive characteristics will be taken, and recorded on the Individual Data Collection Form. Following this, the use of the Facial Expressions Pain Rating Scale will be explained to the children in simple language that they can understand. Peripheral intravenous catheterization will be performed by an experienced nurse working in the pediatric emergency service who is involved in the research. A number 24 peripheral intravenous catheter will be used with all of the pediatric patients. Children in whom the entry to the vein is unsuccessful will not be included in the study. Peripheral intravenous catheterization will be implemented on the veins of either the right or the left arm. The procedural steps of the standard vein entry protocol will be followed with all of the children in the implementation and control groups.

In addition to the standard vein entry protocol, the following interventions will be conducted with the pediatric patients in the implementation groups.

Peripheral intravenous catheterization with pediatric patients in the Buzzy® group: From one minute before the location of the catheter and until the end of the procedure, the researchers will place the Buzzy® device approximately 5cm above the area where the procedure will take place, with its wings under it. The gel in its wings will have been previously frozen solid in a refrigerator. In this way, vibration and cold will be applied, and immediately afterwards, vein entry will be performed. (For the children's safety, a piece of thin sterile gauze will be placed on the area in order to prevent direct contact between the ice wings and the skin.)

Peripheral intravenous catheterization with pediatric patients in the AccuVein® group: In this group, the veins in the area where the entry is to be performed will be visualized with the AccuVein® infrared vein visualization device, and the standard catheter implementation will be performed in the vein which is decided on for entry.

Peripheral intravenous catheterization with pediatric patients in the control group: With the pediatric patients in the control group, no intervention will be performed before or during the procedure, and routine IV catheterization will be carried out without the use of any device.

Immediately after the procedure has been performed, an assistant researcher who is unaware of the catheterization method used will ask the children of all groups to assess their pain levels with the Facial Expressions Pain Rating Scale, and the scores indicated will be recorded on the data collection form. While the study is being conducted, the necessary measures will be taken to prevent the children included in the study from influencing each other, such as not allowing them to see the method applied to the other children.

ELIGIBILITY:
Inclusion Criteria:

* Being aged 7-12 years
* Themselves and their parents participating voluntarily in the study
* Being able to correctly evaluate the Facial Expressions Pain Rating Scale
* Not having, in the area or extremity in which the implementation will be conducted, anything which could interfere with the intervention, such as symptoms or signs of infection, scar tissue, vein or nerve damage or loss of sensation
* Not having used an analgesic in the previous six hours
* Being able to speak and understand Turkish
* Having no visual, auditory or speaking problems
* Not having any condition which could affect the sensation of pain
* Having a peripheral intravenous catheter for the first time in the emergency service

Exclusion Criteria:

* Being mentally retarded
* Having a chronic or fatal illness
* Having any psychiatric diagnosis
* Being unconscious or being unable to communicate verbally
* Not having a vein opened for the first time
* Agitation in themselves or their family
* Themselves or their parents not wanting to participate in the study, or wishing to withdraw at some point during the study
* Any situation which could affect the sensation of pain
* Being younger than seven or older than 12 years

Ages: 7 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 90 (Estimated)
Dates: Start 2022-08-31 (Estimated); Primary Completion 2022-11-10 (Estimated); Study Completion 2022-11-20 (Estimated)

PRIMARY OUTCOMES:
Pain Scores on the Facial Expressions Pain Rating Scale | 4 months
  pain severity in mm
  (Immediately after the procedure has been performed, an assistant researcher will ask the children of all groups to assess their pain severity with the Facial Expressions Pain Rating Scale, and the scores indicated will be recorded on the data collection form)

SECONDARY OUTCOMES:
weight | 4 months
  weight in kilograms
height | 4 months
  height in meters
body mass index (BMI) | 4 months
  BMI in kg/m^2
duration of catheterization | 4 months
  duration of catheterization in second

CONTACTS AND LOCATIONS:
Overall Officials: Seçil Salarcı, MSc, Study Chair — Pediatric Emergency Service of the Health Research and Application Center of Bursa Uludağ University

IPD SHARING:
Plan to Share IPD: No